CLINICAL TRIAL: NCT02442843
Title: Non-invasive Brain Stimulation for Post-Traumatic Stress Disorder
Brief Title: Non Invasive Brain Stimulation for PTSD
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Benjamin Hampstead, PhD, Investigator, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00089481; 1R21MH102539-01 (NIH)
Record Dates: First submitted 2015-02-17; First posted 2015-05-13 (Estimated); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Posttraumatic Stress Disorder (PTSD)
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- active tDCS (Experimental): Investigators will use cathodal tDCS to inhibit the brain regions that may be associated with symptoms of PTSD (temporal cortex). Active tDCS will be provided at 2 miliamps (mA) for 20 minutes (with gradual increase and withdraw of stimulation during the first and last minute).
  Interventions: Device: Active tDCS
- sham tDCS (Sham Comparator): Participants randomized to the sham condition will receive stimulation during the first and final minutes of the 20 minute period (with gradual increase and removal of current during that time).
  Interventions: Device: Sham tDCS
- Combat Controls (No Intervention): Participants without PTSD will undergo neuropsychological testing and a single fMRI scan.

INTERVENTIONS:
Device: Active tDCS — Participants will be randomized into active or sham stimulation in the first tDCS session. Participants will then have the option to complete 9 additional session of tDCS which will be active tDCS or a combination of active and sham tDCS in a non-randomized manner over two consecutive weeks. Each session will last 1 - 2 hours.
  Other Names: mild brain stimulation; HD-tDCS
  Arms: active tDCS
Device: Sham tDCS — Participants will be randomized into active or sham stimulation in the first tDCS session. Participants will then have the option to complete 9 additional session of tDCS which will be active tDCS or a combination of active and sham tDCS in a non-randomized manner over two consecutive weeks. Each session will last 1 - 2 hours.
  Other Names: fake tDCS
  Arms: sham tDCS

SUMMARY:
This study is designed to identify changes in the brain that underlie symptoms of combat-related PTSD using brain imaging (fMRI). Then, the investigators will administer mild electrical stimulation to the side of the head (using a method called tDCS) in an attempt to reduce the symptoms of PTSD.

DETAILED DESCRIPTION:
Being involved in combat is a horrific experience that substantially increases the risk of developing posttraumatic stress disorder (PTSD). Although several effective treatments have been identified for PTSD a substantial number of patients (up to 50%) continue to experience symptoms. The field of neuroscience has revealed that patients with PTSD demonstrate altered functioning within, and interactions between, several brain regions; findings that are consistent with animal models of chronic stress. Despite this evidence, existing treatments are generally not designed using this neuroanatomical knowledge. The central premise of the proposed study is that neuroscientifically-based information can be used to develop more precise and effective treatments. Transcranial direct current stimulation (tDCS) will be used in an attempt to "correct" the dysfunctional brain regions (and communication between these regions), with the expectation that this modulation will result in symptom improvement.

The primary goals of the study are to verify the maladaptive brain networks and then establish evidence that tDCS modulates these networks. Subsequent studies, performed during the later study years, will examine dose-response relationships and synergistic effects of tDCS and existing treatments. Outcome will be assessed using a multi-method approach that includes functional connectivity using resting-state functional magnetic resonance imaging data, neuropsychological tests, and self-report measures of emotional functioning. The combined results will provide vital methodological, mechanistic, and practical information necessary for a formal clinical trial of tDCS in PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Combat Veteran - both Veterans with and without PTSD will be included at different points in this study
* Right-handed
* Between the ages 18-88
* Stable on medications for a minimum of 2 weeks

Exclusion Criteria:

1. a history of neurological disease (e.g., dementia, epilepsy, stroke, moderate - severe traumatic brain injury)
2. "severe" Axis I diagnoses (e.g., bipolar disorder, schizophrenia)
3. presence of Axis II disorders
4. current alcohol or drug abuse/dependence (in the past 8 weeks)
5. participants will also be excluded if they are not MRI compatible (assessed using the guidelines of the American College of Radiology)
6. Imminent risk of harm to self or others
7. history of HIV or sickle cell anemia, as these can cause neuropsychological issues .

Ages: 18 Years to 88 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Functional Connectivity changes as assessed by fMRI images | Pre and post tDCS; typically within 4 weeks
  Investigators will use the fMRI images taken from before and after tDCS to determine if the treatment intervention contributed to any changes within the neural networks associated with the symptoms of PTSD.

SECONDARY OUTCOMES:
Symptomatic changes as assessed by structured questionnaires (PCL-C) | Pre and post tDCS; typically within 4 weeks
  PTSD checklist
Symptomatic changes as assessed by structured questionnaires (CAPS) | Pre and post tDCS; typically within 4 weeks
  Clinician administered PTSD Scale
Symptomatic changes as assessed by structured questionnaires (Hamilton Depression Rating Scale) | Pre and post tDCS; typically within 4 weeks
  Current symptoms of depression
Symptomatic changes as assessed by structured questionnaires (State-trait anxiety inventory) | Pre and post tDCS; typically within 4 weeks
  current symptoms of anxiety
Cognitive changes as assessed by Neuropsychological testing | Pre and post tDCS; typically within 4 weeks
  Verbal (HVLT) and visuospatial memory (object-location association test)
Cognitive changes as assessed by Neuropsychological testing | Pre and post tDCS; typically within 4 weeks
  Working memory (n-back)
Cognitive changes as assessed by Neuropsychological testing | Pre and post tDCS; typically within 4 weeks
  inhibitory control (go/no-go; flanker task; pattern comparison task)
Cognitive changes as assessed by Neuropsychological testing | Pre and post tDCS; typically within 4 weeks
  Executive functioning (Dimensional change card sort)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Hampstead, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Neuropsychology Section, Ann Arbor, Michigan, United States